CLINICAL TRIAL: NCT04572581
Title: Use of Human Milk-Based Diet in the Late Preterm and Term Infant in the Neonatal Intensive Care Unit: A Pilot Randomized Controlled Trial
Brief Title: Donor Breast Milk and Breastfeeding Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Kara L. Calkins, MD, Health Sciences Clinical Assistant Professor, Pediatric Neonatology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-002179
Record Dates: First submitted 2020-09-15; First posted 2020-10-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Breastfeeding, Exclusive; Breastfeeding
Keywords: Late Preterm; Donor Breast Milk
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exclusively Human Milk Diet (Experimental): This group will receive human milk only. If the mother is not producing enough breast milk, this group will receive donor milk supplementation.
  Interventions: Other: Donor Breast Milk
- Formula-based Diet (No Intervention): If the mother is not producing enough breast milk, this group will receive formula supplementation (the standard of care).

INTERVENTIONS:
Other: Donor Breast Milk — Donor breast milk will be given to the newborn if supplementation is required
  Arms: Exclusively Human Milk Diet

SUMMARY:
The purpose of this pilot study is to determine if a randomized controlled study comparing a human milk diet versus a formula supplemented diet in late preterm and term infants in the neonatal intensive care unit (NICU) is feasible.

DETAILED DESCRIPTION:
In late preterm infants and term neonates in the NICU whose mothers intend to breastfeed, this pilot study seeks to 1. determine study feasibility (consent rate, study completion rate, and rate of adherence to study diet), and 2. determine whether a dietary supplementation with donor human milk vs. formula improves: a. the percentage of maternal milk consumption at time of discharge from the NICU, or 7 days of age, whichever is later, b. breastfeeding rates and intent to breastfeed at 6-8 weeks chronological age, and c. breast feeding duration.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age >34 weeks and 0 days
* Mother's intent to breast feed
* NICU admission which is predicted to be at least 72 hours from time of admission

Exclusion Criteria:

* Confirmed genetic disorders and syndromes or other disorders known to affect growth and ability to bottle feed or breast feed (i.e., Trisomies)
* Common neonatal congenital anomalies (cardiac disease, congenital gastrointestinal disorders, etc)
* Commonly accepted contraindications for breast feeding (HIV, galactosemia, herpes lesions on the breast, maternal use of drugs that are considered contraindicated with breast feeding including marijuana)
* Infant admitted to the intensive care unit who is receiving invasive respiratory support (intubation) and/or ionotropic medications
* Any infant whose care is considered futile by the primary medical team

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-06-26 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Study Feasibility_1 | 6-8 weeks chronological age
  Feasibility will be evaluated by: consent rate
Study Feasibility_2 | 6-8 weeks chronological age
  Feasibility will be evaluated by: study completion rate
Study Feasibility_3 | 6-8 weeks chronological age
  Feasibility will be evaluated by: rate of adherence to the study diet.

SECONDARY OUTCOMES:
Percentage of Human Milk Consumption at Discharge | at the time of NICU discharge or 7 days of age, whichever is later
  Maternal milk/total milk (percent) consumed by the neonate over 48 hours
Percentage of Human Milk Consumption After Discharge | 6-8 weeks chronological age
  Maternal milk/total milk (percent) consumed by the infant over 48 hours
Breastfeeding duration | 6-8 weeks chronological age
  time infant received breastmilk since birth
Intent to Breastfeed | 6-8 weeks chronological age
  Mother's desire to continue to breastfeed: specifically assessed by asking the mother if she plans to exclusively breastfeed or not. Answers will be recorded as yes or no.
Growth: Weight | 6-8 weeks chronological age
  Weight in kilograms reported as a z-score
Growth: Height | 6-8 weeks chronological age
  height in centimeters reported as a z-score
Growth: Head Circumference | 6-8 weeks chronological age
  head circumference in centimeters reported as a z-score

OTHER OUTCOMES:
Intestinal Microbiome: microbial profiling (genus level) | 7 days of age
  Microbial profiling (genus level) will be investigated by sequencing of the V4 region of the 16S ribosomal ribonucleic acid gene
Intestinal Microbiome: alpha diversity (Chao1) | 7 days of age
  Alpha diversity (Chao1) will be investigated by sequencing of the V4 region of the 16S ribosomal ribonucleic acid gene

CONTACTS AND LOCATIONS:
Overall Officials: Kara L Calkins, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Santa Monica-UCLA, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No
There is no current plan to make IPD available for other research given this is a small pilot feasibility study.

REFERENCES:
- [Background] Adamkin DH. Feeding problems in the late preterm infant. Clin Perinatol. 2006 Dec;33(4):831-7; abstract ix. doi: 10.1016/j.clp.2006.09.003. PMID 17148007
- [Background] Agostoni C, Buonocore G, Carnielli VP, De Curtis M, Darmaun D, Decsi T, Domellof M, Embleton ND, Fusch C, Genzel-Boroviczeny O, Goulet O, Kalhan SC, Kolacek S, Koletzko B, Lapillonne A, Mihatsch W, Moreno L, Neu J, Poindexter B, Puntis J, Putet G, Rigo J, Riskin A, Salle B, Sauer P, Shamir R, Szajewska H, Thureen P, Turck D, van Goudoever JB, Ziegler EE; ESPGHAN Committee on Nutrition. Enteral nutrient supply for preterm infants: commentary from the European Society of Paediatric Gastroenterology, Hepatology and Nutrition Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2010 Jan;50(1):85-91. doi: 10.1097/MPG.0b013e3181adaee0. PMID 19881390
- [Background] Backstrom MC, Aine L, Maki R, Kuusela AL, Sievanen H, Koivisto AM, Ikonen RS, Maki M. Maturation of primary and permanent teeth in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2000 Sep;83(2):F104-8. doi: 10.1136/fn.83.2.f104. PMID 10952702
- [Background] Cleaveland K. Feeding challenges in the late preterm infant. Neonatal Netw. 2010 Jan-Feb;29(1):37-41. doi: 10.1891/0730-0832.29.1.37. PMID 20085875
- [Background] Darcy AE. Complications of the late preterm infant. J Perinat Neonatal Nurs. 2009 Jan-Mar;23(1):78-86. doi: 10.1097/JPN.0b013e31819685b6. PMID 19209064
- [Background] DeMauro SB, Patel PR, Medoff-Cooper B, Posencheg M, Abbasi S. Postdischarge feeding patterns in early- and late-preterm infants. Clin Pediatr (Phila). 2011 Oct;50(10):957-62. doi: 10.1177/0009922811409028. Epub 2011 Aug 19. PMID 21856965
- [Background] Engle WA, Tomashek KM, Wallman C; Committee on Fetus and Newborn, American Academy of Pediatrics. "Late-preterm" infants: a population at risk. Pediatrics. 2007 Dec;120(6):1390-401. doi: 10.1542/peds.2007-2952. PMID 18055691
- [Background] Fein SB, Labiner-Wolfe J, Shealy KR, Li R, Chen J, Grummer-Strawn LM. Infant Feeding Practices Study II: study methods. Pediatrics. 2008 Oct;122 Suppl 2:S28-35. doi: 10.1542/peds.2008-1315c. PMID 18829828
- [Background] Gauer RL, Burket J, Horowitz E. Common questions about outpatient care of premature infants. Am Fam Physician. 2014 Aug 15;90(4):244-51. PMID 25250998
- [Background] Gianni ML, Bezze EN, Sannino P, Baro M, Roggero P, Muscolo S, Plevani L, Mosca F. Maternal views on facilitators of and barriers to breastfeeding preterm infants. BMC Pediatr. 2018 Aug 27;18(1):283. doi: 10.1186/s12887-018-1260-2. PMID 30149811
- [Background] Jain BK. Vitamin requirements of very low birth weight infants: a review. Indian J Matern Child Health. 1994 Apr-Jun;5(2):46-9. PMID 12318806
- [Background] Kalyoncu O, Aygun C, Cetinoglu E, Kucukoduk S. Neonatal morbidity and mortality of late-preterm babies. J Matern Fetal Neonatal Med. 2010 Jul;23(7):607-12. doi: 10.1080/14767050903229622. PMID 19757335
- [Background] Lapillonne A, O'Connor DL, Wang D, Rigo J. Nutritional recommendations for the late-preterm infant and the preterm infant after hospital discharge. J Pediatr. 2013 Mar;162(3 Suppl):S90-100. doi: 10.1016/j.jpeds.2012.11.058. PMID 23445854
- [Background] Lucas A, Morley R, Cole TJ, Gore SM. A randomised multicentre study of human milk versus formula and later development in preterm infants. Arch Dis Child Fetal Neonatal Ed. 1994 Mar;70(2):F141-6. doi: 10.1136/fn.70.2.f141. PMID 8154907
- [Background] Lucas A, Morley R, Cole TJ. Randomised trial of early diet in preterm babies and later intelligence quotient. BMJ. 1998 Nov 28;317(7171):1481-7. doi: 10.1136/bmj.317.7171.1481. PMID 9831573
- [Background] Meier P, Patel AL, Wright K, Engstrom JL. Management of breastfeeding during and after the maternity hospitalization for late preterm infants. Clin Perinatol. 2013 Dec;40(4):689-705. doi: 10.1016/j.clp.2013.07.014. Epub 2013 Sep 21. PMID 24182956
- [Background] Raju TN, Higgins RD, Stark AR, Leveno KJ. Optimizing care and outcome for late-preterm (near-term) infants: a summary of the workshop sponsored by the National Institute of Child Health and Human Development. Pediatrics. 2006 Sep;118(3):1207-14. doi: 10.1542/peds.2006-0018. PMID 16951017
- [Background] Raju TN. Late-preterm births: challenges and opportunities. Pediatrics. 2008 Feb;121(2):402-3. doi: 10.1542/peds.2007-2357. No abstract available. PMID 18245431
- [Background] Schanler RJ, Shulman RJ, Lau C. Feeding strategies for premature infants: beneficial outcomes of feeding fortified human milk versus preterm formula. Pediatrics. 1999 Jun;103(6 Pt 1):1150-7. doi: 10.1542/peds.103.6.1150. PMID 10353922
- [Background] Schanler RJ, Lau C, Hurst NM, Smith EO. Randomized trial of donor human milk versus preterm formula as substitutes for mothers' own milk in the feeding of extremely premature infants. Pediatrics. 2005 Aug;116(2):400-6. doi: 10.1542/peds.2004-1974. PMID 16061595
- [Background] Tomashek KM, Shapiro-Mendoza CK, Weiss J, Kotelchuck M, Barfield W, Evans S, Naninni A, Declercq E. Early discharge among late preterm and term newborns and risk of neonatal morbidity. Semin Perinatol. 2006 Apr;30(2):61-8. doi: 10.1053/j.semperi.2006.02.003. PMID 16731278
- [Background] Torrazza RM, Neu J. The altered gut microbiome and necrotizing enterocolitis. Clin Perinatol. 2013 Mar;40(1):93-108. doi: 10.1016/j.clp.2012.12.009. PMID 23415266
- [Background] Giapros VI, Schiza V, Challa AS, Cholevas VK, Theocharis PD, Kolios G, Pantou C, Andronikou SK. Vitamin D and parathormone levels of late-preterm formula fed infants during the first year of life. Eur J Clin Nutr. 2012 Feb;66(2):224-30. doi: 10.1038/ejcn.2011.158. Epub 2011 Sep 7. PMID 21897423
- [Background] Ip S, Chung M, Raman G, Trikalinos TA, Lau J. A summary of the Agency for Healthcare Research and Quality's evidence report on breastfeeding in developed countries. Breastfeed Med. 2009 Oct;4 Suppl 1:S17-30. doi: 10.1089/bfm.2009.0050. PMID 19827919
- [Background] Valentine G, Chu DM, Stewart CJ, Aagaard KM. Relationships Between Perinatal Interventions, Maternal-Infant Microbiomes, and Neonatal Outcomes. Clin Perinatol. 2018 Jun;45(2):339-355. doi: 10.1016/j.clp.2018.01.008. Epub 2018 Feb 23. PMID 29747892
- [Background] Walker M. Breastfeeding the late preterm infant. J Obstet Gynecol Neonatal Nurs. 2008 Nov-Dec;37(6):692-701. doi: 10.1111/j.1552-6909.2008.00293.x. PMID 19012718
- [Background] Young L, Morgan J, McCormick FM, McGuire W. Nutrient-enriched formula versus standard term formula for preterm infants following hospital discharge. Cochrane Database Syst Rev. 2012 Mar 14;(3):CD004696. doi: 10.1002/14651858.CD004696.pub4. PMID 22419297
- [Background] Caporaso JG, Lauber CL, Walters WA, Berg-Lyons D, Huntley J, Fierer N, Owens SM, Betley J, Fraser L, Bauer M, Gormley N, Gilbert JA, Smith G, Knight R. Ultra-high-throughput microbial community analysis on the Illumina HiSeq and MiSeq platforms. ISME J. 2012 Aug;6(8):1621-4. doi: 10.1038/ismej.2012.8. Epub 2012 Mar 8. PMID 22402401
- [Background] Callahan BJ, McMurdie PJ, Rosen MJ, Han AW, Johnson AJ, Holmes SP. DADA2: High-resolution sample inference from Illumina amplicon data. Nat Methods. 2016 Jul;13(7):581-3. doi: 10.1038/nmeth.3869. Epub 2016 May 23. PMID 27214047